CLINICAL TRIAL: NCT02812810
Title: Evaluation of the Efficacy of Low-frequency rTMS on Craving in Smoking Dependence: Single-centre Randomized, Controlled Blinded Pilot Study
Brief Title: Evaluation of the Efficacy of Repetitive Transcranial Magnetic Stimulation (rTMS) Low-frequency on Craving in Smoking Dependence
Acronym: rTMS TABAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TROJAK DRCI 2010
Record Dates: First submitted 2016-06-20; First posted 2016-06-24 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Smoking Cessation; Addiction
MeSH Terms: conditions — Smoking Cessation; Behavior, Addictive

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- active rTMS (Experimental)
  Interventions: Device: active rTMS
- placebo rTMS (Placebo Comparator)
  Interventions: Device: sham rTMS

INTERVENTIONS:
Device: active rTMS
  Arms: active rTMS
Device: sham rTMS
  Arms: placebo rTMS

SUMMARY:
The fight against smoking is a public health priority. Without help, fewer than 5% of des smokers are abstinent at 12 months after smoking cessation.

Despite well-managed attempts at smoking cessation with nicotine substitutes, the rate of success at 12 months in patients dependent on nicotine is only 18%. Moreover, other therapeutic strategies (acupuncture, hypnosis…) have not proved to be effective.

The investigators propose a new therapeutic strategy for smoking cessation, which is based on associating nicotine substitutes (to reduce physical symptoms of weaning from nicotine) with rTMS at 1 Hz to the right DorsoLateral PreFrontal Cortex (DLPFC) for 2 weeks (to diminish craving for tobacco). The principal objective is to improve the success rate for smoking cessation attempts in patients who are highly dependent on nicotine, and who have failed using usual smoking cessation strategies.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18-65 years old
* Wishing to stop smoking
* Highly dependent on nicotine (score ≥ 7 on the Fagerström self-questionnaire)
* History of at least 2 failed attempts to stop smoking despite recommended treatments (nicotine, vareniciline, bupropion)

Exclusion Criteria:

* Abstinence in the 3 previous months
* Absence of effective contraception for women
* Progressive chronic disease
* Ongoing psychiatric disorders
* Current addiction to other substances or cessation of less than one year
* Current treatment with psychotropic agents
* Epilepsy and other contra-indications for rTMS (pacemaker, metallic clips or other electronic implants, head trauma, intracranial hypertension).
* Contra-indications for transdermal nicotine substitutes (recent myocardial infarction, unstable or worsening angina, Prinzmetal angina, severe heart rhythm disorders, recent stroke, skin disorders that could interfere with the use of transdermal treatments, hypersensitivity to one of the constituents).
* Personnel working in the psychiatric and addictology unit of the CHU (conflict of interest)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-09; Primary Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline score of Tabacco Craving Questionnaire (TCQ) | at Week 0, Week 1, Week 2, Week 6 and Week 12 after stimulation

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire, Dijon, France

REFERENCES:
- [Result] Trojak B, Meille V, Achab S, Lalanne L, Poquet H, Ponavoy E, Blaise E, Bonin B, Chauvet-Gelinier JC. Transcranial Magnetic Stimulation Combined With Nicotine Replacement Therapy for Smoking Cessation: A Randomized Controlled Trial. Brain Stimul. 2015 Nov-Dec;8(6):1168-74. doi: 10.1016/j.brs.2015.06.004. Epub 2015 Jun 16. PMID 26590478